CLINICAL TRIAL: NCT06001749
Title: Feasibility Phase 2 Study of Psilocybin-Assisted Therapy for Opioid-Refractory Pain in Patients With Advanced Cancer
Brief Title: Psilocybin in Cancer Pain Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yvan Beaussant, MD, MSci (Other)
Collaborators: Cy Biopharma (Unknown); Pancreatic Cancer North America (Unknown)
Responsible Party: Sponsor-Investigator, Yvan Beaussant, MD, MSci, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-325
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Opioid-Related Disorders; Pain Management; Pain Management and Care; Advanced Cancer; Advanced Cancers
Keywords: Opioid-Related Disorders; Pain Management; Pain Management and Care; Advanced Cancer; Advanced Cancers
MeSH Terms: conditions — Opioid-Related Disorders; Agnosia | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): Participants will complete study procedures as follows:
  * 2, in-clinic or remote, preparation sessions with therapists.
  * In-clinic treatment session with therapists at Dana-Farber Cancer Institute. Participants will take a predetermined amount of psilocybin once. Participants will be transported home by a friend or family member.
  * In-clinic integration session the day after psilocybin administration with therapists.
  * In-clinic or remote, integration session with therapists 1 week after psilocybin administration.
  * In-clinic or remote follow visits with therapists at week 2, 3, 5, 8, and 12 after psilocybin administration.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — A tryptamine derivative, capsule, taken orally.

SUMMARY:
The overall objective of this study is to assess the feasibility, safety and preliminary efficacy of psilocybin-assisted therapy to alleviate opioid-refractory pain in patients with advanced-cancer.

The name of the study intervention used in this research study is:

Psilocybin (a tryptamine derivative)

DETAILED DESCRIPTION:
This study is a phase 2 open label, single center, concurrent mixed-methods trial to assess the feasibility of a novel palliative-care informed psilocybin-assisted psychotherapy regimen to alleviate opioid-refractory pain in patients with advanced-cancer. Psilocybin works on the serotonin system in the brain which is linked to the regulation of mood, motivation and impulse control.

Psilocybin is an "Investigational" drug, meaning that the study drug has not been approved by the U.S. Food and Drug Administration (FDA) as a treatment for any disease. However, investigators have permission from the FDA to use this drug in this research study.

The research study procedures include screening for eligibility, an electrocardiogram, blood tests, and the study intervention includes preparation, evaluations, one psilocybin session and follow up visits.

Participants will be followed for up to 12 weeks (approximately 3 months) after receiving the study treatment.

It is expected that about 15 people will take part in this research study.

Filament Health is supporting this research study by providing the study investigational medication, psilocybin.

Cy Biopharma and Pancreatic Cancer North America are supporting this research study by providing funding.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 year old or older;
* Participants must have advanced cancer, defined as a cancer that is unlikely to be cured or controlled with treatment;
* Participants must have progressed on or be intolerant to approved therapies with a known clinical benefit (unless it is documented that they have refused such treatments);
* Participants must evaluate their average pain on BPI Severity Scale ≥ 4/10 over the past week;
* Participants must receive chronic opioid pharmacotherapy for pain with an Oral Morphine Equivalent (OME) ≥ 200mg/day;
* Participants must have been seen by a palliative care clinician either at DFCI, MGH or associated satellites in the last three months;
* Participants must have an ECOG Performance Status ≤ 2
* Participants must meet the following organ and marrow function on their last available bloodwork as defined below:

  * Platelets ≥ 50,000/mcL
  * AST(SGOT)/ALT(SGPT) ≤ 5 × institutional ULN
* Participants must be able to understand and willing to sign a written informed consent document
* Participants must be able to swallow pills.
* Participants must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
* Participants must agree to inform the investigators within 48 hours of any new medical conditions and procedures.
* Participants must agree to the following lifestyle modifications (described in more detail in Section 3.4 Lifestyle Modifications):

  * Comply with requirements for diet,
  * Refrain from certain medications prior to Experimental Sessions,
  * Be driven home after each Experimental Session,
  * Commit to medication dosing, therapy, and study procedures.

Exclusion Criteria:

* Participants who receive concurrent (less than four weeks or planned within 6 weeks) cytotoxic chemotherapy or radiation therapy that may impair general level of physical functioning or affect study outcomes;
* Participants with a condition impairing oral intake or digestive absorption;
* Participants who are not able to give adequate informed consent;
* Participants who have a significant suicide risk as defined by suicidal ideation with intent and with or without a plan as endorsed on items 4 and/or 5 on the C-SSRS within the past 6 months or at V0
* Participants who have a history of, or a current diagnostic of primary psychotic disorder, major depressive disorder with psychotic features, bipolar affective disorder type 1 or history of or current dissociative identity disorder; and participants who have an ongoing substance use disorder (defined as active in the past year). Participants with first-degree relatives with schizophrenia or bipolar disorder may be eligible depending on their age and personal and family psychiatric history. The decision will be made by the principal investigator and study psychiatrist based on risk assessment.
* Participants for whom there is a potential for adverse drug-drug interactions. Concomitant medications with significant potential to interact with study medications will be exclusionary if they cannot be tapered. These include the following:

  * Serotoninergic antidepressants
  * Serotonin and Norepinephrine Reuptake Inhibitors (SNRIs)
  * Tricyclic Antidepressants (TCAs)
  * Efavirenz
  * serotonin-acting dietary supplements (i.e. 5-hydroxy-tryptophan or St. John's wort)
  * Centrally-acting serotonergic agents (e.g. MAO inhibitors)
  * Antipsychotics (e.g. first and second generation)
  * Mood stabilizers (e.g. lithium, valproic acid)
  * Aldehyde dehydrogenase inhibitors (e.g. disulfiram)
  * Significant inhibitors of UGT 1A0 or UGT 1A10 Any psychiatric medication will be tapered if possible in an appropriate fashion to avoid withdrawal effects. They will be discontinued long enough before the psilocybin Session to avoid the possibility of any drug-drug interaction (the interval will be at least five times the particular drug and active metabolites' half-life + one week for stabilization). See section 5.3 of the protocol for concomitant medications and tapering instructions.
* Participants who have evidence or history of significant (controlled or uncontrolled) hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder, or any other medical disorder judged by the investigator to significantly increase the risk of psilocybin administration (participants with hypothyroidism who are on adequate and stable thyroid replacement will not be excluded).
* Participants with brain tumors or brain metastases that haven't been successfully treated
* Participants with lab abnormalities that may contribute to somnolence, confusion or delayed metabolism of psilocybin and/or with severe lab abnormalities (grade 3 or more per CTCAE scale).
* Participants with a diagnosis of cirrhosis or liver failure
* Participants who have uncontrolled hypertension using the standard criteria of the American Heart Association (values of 140/90 milligrams of Mercury [mmHg] or higher assessed on three separate occasions)
* Participants who have a heart rate > 100 bpm on three separate occasions
* Participants who have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease.
* Participants who have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
* Participants who have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening. Participants with a history of atrial fibrillation, atrial tachycardia, atrial flutter or paroxysmal supraventricular tachycardia or any other arrhythmia associated with a bypass tract may be enrolled if they have been successfully treated.
* Participants who have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Participants who have a history of myocardial infarction, coronary artery disease or heart failure
* Participants who have a marked Baseline prolongation of QT/QTc interval. For purposes of eligibility, this is defined as repeated demonstration of a QT interval corrected on the triplicate ECGs performed at screening, using Fridericia's formula [QTcF] > 450 milliseconds [ms] in males and > 460 ms in females.
* For transgender or non binary participants, QTc interval will be evaluated based on sex assigned at birth, unless the participant has been on hormonal treatment for five or more years.
* Women who are pregnant, nursing, or able to become pregnant and are not practicing an effective means of birth control. Acceptable methods of contraception are the following: intrauterine device, injected/ implanted/ intravaginal/ transdermal hormonal method, oral hormones plus a barrier contraception, abstinence, vasectomized sole partner, or double barrier contraception.
* Participants who have hypersensitivity to any ingredient of the IMP (Investigational Medicinal Product).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Psilocybin-Assisted Therapy | 3 weeks
  Feasibility of intervention is defined as at least 60% of recruited participants will complete treatment and all assessments.
Acceptability of Psilocybin-Assisted Therapy | 3 weeks
  Acceptability is defined as >= 70% of participants will evaluate favorably (agree or strongly agree) acceptability on the Reactions to Research Participation Questionnaire Revised (RRPQ V6b), a 23-item measure scored on a 5-point Likert scale.

SECONDARY OUTCOMES:
Change in Pain Intensity Score from Baseline | 3 weeks
  Pain intensity score is evaluated by the Brief Pain Inventory (BPI)-short, and change will be calculated between the score at baseline and at assessment at week 3 post dosing. Pain intensity score ranges from 0-10, while a larger number represents worse feelings.
Change in Pain Interference Score from Baseline | 3 weeks
  Pain interference score is evaluated by the Brief Pain Inventory (BPI)-short, and change will be calculated between the score at baseline and at assessment at week 3 post dosing. Pain interference score ranges from 0-10, while a larger number represents worse feelings.
Change in Pain Catastrophizing Score from Baseline | 3 weeks
  Pain catastrophizing is measured by the Pain Catastrophizing Scale (PCS), which consists of 13 items describing different thoughts and feelings associated with catastrophizing response-style. Answers are graded on a 5-point scale with endpoints (0) not at all to (4) all the time.
Change in Oral Morphine Equivalent (OME) from Baseline | 3 weeks
  OME would be obtained from participant's Electronic Medical Record and/or directly from participants based on CDC Oral Morphine Milligram Equivalent Conversion table.

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Beaussant, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu